CLINICAL TRIAL: NCT04554524
Title: Single-Arm Study to Carbo-paclitaxel/ Nab-paclitaxel Combined With Pembrolizumab as the First Line Therapy in Treating Patients With Locally Advanced or Metastatic Invasive Thymoma and Thymic Carcinoma That Cannot Be Removed by Surgery
Brief Title: Chemotherapy Combined With Pembrolizumab in Treating Patients With Thymoma and Thymic Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Yongan Zhou, MD, Chief physician of Thoracic Surgery, Principal Investigator, Tang-Du Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K202008-07
Record Dates: First submitted 2020-09-07; First posted 2020-09-18 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Thymoma and Thymic Carcinoma
Keywords: Thymoma; Thymic carcinoma; Pembrolizumab
MeSH Terms: conditions — Thymoma | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy+Pembrolizumab (Experimental): Chemotherapy combined with pembrolizumab.
  Interventions: Drug: Chemotherapy+Pembrolizumab.

INTERVENTIONS:
Drug: Chemotherapy+Pembrolizumab. — Eligible subjects will receive 4 cycles carbo-paclitaxel/ nab-paclitaxel combined with pembrolizumab. Response rate assessed by the site investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). After 4 cycles treatment, complete response subjects continue carbo-paclitaxel/ nab-paclitaxel combined with pembrolizumab up to disease progression, some of partial disease and stable disease subjects can receive surgical treatment. And then continue carbo-paclitaxel/ nab-paclitaxel combined with pembrolizumab up to disease progression, other partial disease and stable disease subjects cannot be removed by surgery will continue carbo-paclitaxel/ nab-paclitaxel combined with pembrolizumab for 4 cycles and then pembrolizumab or Normal Saline up to disease progression.
  Other Names: Carbo-paclitaxel/ nab-paclitaxel

SUMMARY:
This is an investigational, single arm study.

DETAILED DESCRIPTION:
Pembrolizumab is FDA approved and commercially available for treatment of many types of cancers. It is considered investigational to use chemotherapy combined with pembrolizumab to treat thymoma or Thymic carcinoma.

Subjects will be evaluated for eligibility during a 28-day screening period. Eligible subjects will receive 4 cycles carbo-paclitaxel/ nab-paclitaxel combined with pembrolizumab. Response rate assessed by the site investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).

Up to 40 participants will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of unresectable thymoma or thymic carcinoma.
2. Have measurable disease based on RECIST 1.1.
3. Patients must not have had prior systemic anti-cancer therapy for locally advanced or metastatic unresectable thymoma or thymic carcinoma.
4. Patients who could provision of archival to evaluate the PD-L1 expression status.
5. Be ≥ 18 years of age on day of signing informed consent.
6. Life expectancy > 3 months.
7. Have a performance status (PS) of 0 or 1 on the ECOG PS.
8. Demonstrate adequate organ function as defined below all screening labs should be performed.

   * Hematological: absolute neutrophil count ≥ 1500/mcL; platelets ≥ 80000mcL; hemoglobin ≥ 9g/dL or ≥ 5.6 mmol/L without transfusion within 4 weeks.
   * Renal: serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤ 1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN.
   * Hepatic: serum total bilirubin ≤ 1.5 X ULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN; AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases; albumin ≥ 2.5mg/dL.
   * Coagulation: International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

1. Patients have had prior systemic anti-cancer therapy.
2. Has a known additional malignancy past 5 years. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
3. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 3 days prior to trial treatment.
4. Hypersensitivity to carboplatin or paclitaxel or nab-paclitaxel or any of their excipients.
5. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
6. Asthmatic subjects requiring intermittent use of bronchodilators, inhaled steroids or local steroid injections were not excluded.
7. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent. Participated in any other pembrolizumab trials or was treated with pembrolizumab.
8. Has an active infection requiring systemic therapy.
9. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
10. As known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
11. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate. | After 4 cycles (each cycle is 21 days) treatment up to 4 years.
  Response rate assessed by the site investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Progression-free Survival. | After 4 cycles (each cycle is 21 days) treatment up to 4 years.
  Response rate assessed by the site investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Yongan Zhou, Study Chair — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China